CLINICAL TRIAL: NCT06920667
Title: Effect of a Combined Whey Protein, Creatine, Omega-3, and Vitamin D Supplement on Glycemic Variability in Mexican Patients With Recently Diagnosed Type 2 Diabetes: A Randomized, Double-blind Trial Using Continuous Glucose Monitoring
Brief Title: Effect of a Protein-Creatine-Omega3-Vitamin D Supplement on Glycemic Variability in Mexican Patients With Type 2 Diabetes
Acronym: PROVID-DM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Héctor Iván Saldívar Cerón (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor-Investigator, Héctor Iván Saldívar Cerón, Principal Investigator, Universidad Nacional Autonoma de Mexico
Organization: Universidad Nacional Autonoma de Mexico (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE/FESI/032025/1908; FICDTEM-2023-131 (Other: COMECYT)
Record Dates: First submitted 2025-04-01; First posted 2025-04-10 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Glycemic Variability; Recently Diagnosed Diabetes; Nutrition Intervention; Continuous Glucose Monitoring; Metabolic Biomarkers; Gut Microbiota; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to either a multi-nutrient supplement group or a placebo group. Both arms will follow the same study procedures over a 12-week intervention period, with continuous glucose monitoring and clinical assessments at multiple time points.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a quadruple-blind study. Participants, clinical staff, study investigators, and outcomes assessors will all be blinded to group allocation. Supplement and placebo sachets will be identical in appearance, taste, and packaging, and will be prepared by an external manufacturer (O'HERVANARIO).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supplement Group (Experimental): Participants assigned to this arm will receive a daily nutritional supplement for 12 weeks. The supplement will be provided in powdered sachets containing 30 g of whey protein isolate, 5 g of creatine monohydrate, 1 g of omega-3 fatty acids (EPA/DHA), and 1,000 IU of vitamin D3. Participants will dissolve the sachet in water and consume it once daily. Glycemic variability will be assessed through continuous glucose monitoring at five time points, and clinical evaluations will be performed biweekly.
  Interventions: Dietary Supplement: Protein-Creatine-Omega-3-Vitamin D Supplement
- Placebo Group (Placebo Comparator): Participants in this arm will receive a daily placebo for 12 weeks. The placebo will be formulated with maltodextrin and will be identical in appearance, taste, and packaging to the active supplement. It will not contain whey protein, creatine, omega-3, or vitamin D. Participants will dissolve the sachet in water and consume it once daily. Glycemic variability and all other outcome measures will be assessed in the same schedule and manner as in the intervention group.
  Interventions: Dietary Supplement: Placebo (Maltodextrin)

INTERVENTIONS:
Dietary Supplement: Protein-Creatine-Omega-3-Vitamin D Supplement — Participants will receive a daily powdered supplement containing 30 g of whey protein isolate, 5 g of creatine monohydrate, 1 g of omega-3 fatty acids (EPA/DHA), and 1,000 IU of vitamin D3. The supplement will be taken once daily for 12 weeks, dissolved in water. It is designed to reduce glycemic variability and improve metabolic parameters in individuals with recently diagnosed type 2 diabetes.
  Arms: Supplement Group
Dietary Supplement: Placebo (Maltodextrin) — Participants will receive a daily powdered placebo formulated with maltodextrin, without any active ingredients (no whey protein, creatine, omega-3, or vitamin D). It is identical in appearance, taste, and packaging to the active supplement. It will be taken once daily for 12 weeks and administered in the same conditions as the intervention group.
  Arms: Placebo Group

SUMMARY:
This study aims to evaluate the effect of a daily nutritional supplement containing whey protein, creatine, omega-3 fatty acids, and vitamin D on blood sugar fluctuations in adults with recently diagnosed type 2 diabetes. Forty participants will be enrolled in a 12-week, double-blind, randomized clinical trial. Half of the participants will receive the supplement, while the other half will receive a placebo. Blood sugar levels will be monitored using continuous glucose monitoring (CGM) devices placed at five different time points during and after the intervention. The study will also measure changes in HbA1c, body composition, metabolic biomarkers, and gut microbiota. Participants will receive medical follow-up and support for six months after the study. The goal is to explore whether this supplement can help stabilize glucose levels and support early management of diabetes.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled clinical trial will evaluate the impact of a combined supplement-composed of whey protein, creatine monohydrate, omega-3 fatty acids (EPA/DHA), and vitamin D-on glycemic variability in Mexican adults recently diagnosed with type 2 diabetes (diagnosis within the last 5 years, HbA1c 7.0-10.0%, treated with metformin or no pharmacologic therapy).

Forty participants will be randomized (1:1) to receive either the active supplement or placebo for 12 weeks. Glycemic variability will be assessed through five time points using continuous glucose monitoring (CGM) with FreeStyle Libre sensors. Secondary outcomes include changes in HbA1c, fasting glucose, anthropometric data (via InBody H30), metabolic and inflammatory biomarkers (Bio-Plex Pro Human Diabetes 10-Plex Assay), and gut microbiota composition (via 16S rRNA sequencing in collaboration with the University of Illinois at Chicago).

The study also includes biweekly clinical assessments to monitor adherence and safety, and a final post-intervention follow-up phase four weeks after supplementation ends. All participants will receive six months of free medical follow-up. The study is designed to explore the feasibility of using CGM and multi-nutrient supplementation as part of early, non-pharmacological strategies to improve glycemic control in Latin American populations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Diagnosis of type 2 diabetes mellitus within the past 5 years
* HbA1c between 7.0% and 10.0%
* BMI between 25 and 40 kg/m²
* On metformin monotherapy or no glucose-lowering medications
* Willing to follow study instructions and attend all scheduled visits
* Able to provide written informed consent

Exclusion Criteria:

* Use of insulin or other antidiabetic medications beyond metformin
* History of type 1 diabetes, pancreatitis, or major GI surgery
* Severe renal, hepatic, or cardiovascular disease
* Use of supplements with whey protein, creatine, omega-3, or vitamin D in the past 3 months
* Known allergy to supplement/placebo ingredients
* Participation in another clinical trial within the past 3 months
* Pregnancy or breastfeeding
* Any condition that, in the investigator's judgment, may interfere with study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-10-25 (Estimated)

PRIMARY OUTCOMES:
Change in Glycemic Variability | Baseline, Week 4, Week 8, Week 12, and 4 weeks post-intervention (Week 16)
  Change in Standard Deviation of Glucose Values (mg/dL)
Change in Coefficient of Variation of Glucose (%) | Baseline, Week 4, Week 8, Week 12, and Week 16 (4 weeks post-intervention)
  The coefficient of variation (CV) of glucose levels will be calculated from CGM data to evaluate glycemic variability, reflecting the ratio between the SD and the mean glucose concentration during the monitoring period.
Change in Time in Range (TIR, % of time between 70-180 mg/dL) | Baseline, Week 4, Week 8, Week 12, and Week 16 (4 weeks post-intervention)
  Time in Range (TIR) will be defined as the percentage of time that CGM glucose readings remain within the target range of 70-180 mg/dL. This measure will help assess overall glycemic control during and after the intervention.

SECONDARY OUTCOMES:
Change in Hemoglobin A1c (HbA1c) | Baseline and Week 12
  Glycated hemoglobin (HbA1c) levels will be measured at baseline and post-intervention to assess long-term glycemic control.
Change in Total Fat Mass (kg) | Baseline and Week 12
  Total fat mass will be measured by bioelectrical impedance analysis (BIA) using the InBody H30 device. The change in fat mass in kilograms will be evaluated from baseline to Week 12 to assess the effect of the intervention on body composition.
Change in Metabolic and Inflammatory Biomarkers | Baseline, Week 12
  Plasma levels of selected biomarkers (e.g., insulin, adiponectin, leptin, IL-6, TNF-α) will be measured using Bio-Plex Pro Human Diabetes 10-Plex Assay.
Change in Gut Microbiota Composition | Baseline and Week 12
  Microbiota diversity and relative abundance will be assessed by 16S rRNA sequencing of stool samples.
Change in Skeletal Muscle Mass (kg) | Baseline and Week 12
  Skeletal muscle mass will be assessed via bioelectrical impedance analysis using the InBody H30. The difference in muscle mass from baseline to Week 12 will reflect changes in lean tissue due to the intervention.
Change in Visceral Fat Area (cm²) | Baseline and Week 12
  Visceral fat area will be calculated using the InBody H30 bioimpedance analyzer. The change in cm² from baseline to Week 12 will be used to evaluate the effect of the supplement on abdominal fat.
Change in Plasma Insulin Levels (μIU/mL) | Baseline and Week 12
  Plasma insulin concentrations will be measured using the Bio-Plex Pro Human Diabetes 10-Plex Assay. The change from baseline to Week 12 will help evaluate insulin sensitivity and pancreatic function.
Change in Plasma Adiponectin Levels (μg/mL) | Baseline and Week 12
  Plasma adiponectin levels will be determined using a multiplex assay to assess anti-inflammatory and insulin-sensitizing effects. Changes from baseline to Week 12 will be compared between groups.
Change in Plasma Leptin Levels (ng/mL) | Baseline and Week 12
  Leptin concentrations will be assessed in plasma using the Bio-Plex platform to evaluate changes in energy balance and adipose tissue signaling during the intervention.
Change in Plasma IL-6 Levels (pg/mL) | Baseline and Week 12
  Plasma levels of interleukin-6 (IL-6), a key inflammatory cytokine, will be measured to assess systemic inflammation. The change between baseline and Week 12 will be used as an indicator of intervention impact.
Change in Plasma TNF-α Levels (pg/mL) | Baseline and Week 12
  Plasma tumor necrosis factor alpha (TNF-α) will be quantified to evaluate pro-inflammatory status. The change from baseline to Week 12 will indicate potential anti-inflammatory effects of the intervention.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) to be shared will include baseline and post-intervention values of glycemic variability (CGM metrics), HbA1c, fasting glucose, anthropometric data (body composition, grip strength), inflammatory and metabolic biomarkers, and gut microbiota profiles.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be made available beginning 6 months after publication of the main results and will remain available for 5 years, or until depletion of data access capacity.
Access Criteria: Access will be granted to qualified researchers affiliated with academic or health institutions, upon submission of a methodologically sound proposal. Requests will be reviewed by the principal investigator and ethics committee. Data will be shared through secure institutional platforms or upon direct contact with the research team.